CLINICAL TRIAL: NCT00252330
Title: An Eight-Week, Double-Blind, Placebo Controlled, Multicenter Study With Escitalopram (10 mg qd) as Positive Control, Evaluating the Efficacy, Safety, Tolerability of a Fixed Dose of SR58611A (350 mg q12) in Outpatients With MDD
Brief Title: Efficacy and Safety of SR58611A in Patients With Major Depressive Disorder
Acronym: PHOENIX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5116
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; depression; major depressive episode; antidepressive agents
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Amibegron hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR58611A

SUMMARY:
To evaluate the efficacy of a fixed dose of SR58611A(350 mg q12) compared to placebo in patients with MajorDepressive Disorder (MDD) using escitalopram (10 mgqd) as positive control. In addition, the tolerability and safety of SR58611A in patients with MDD will be evaluated.

DETAILED DESCRIPTION:
To evaluate the efficacy of a fixed dose of SR58611A(350 mg q12) compared to placebo in patients with MajorDepressive Disorder (MDD) using escitalopram (10 mgqd) as positive control. In addition, the tolerability and safety of SR58611A in patients with MDD will be evaluated. The present study is an 8-week, double-blind, placebo- and escitalopram-controlled, randomized, parallel-group study. A 1-week, placebo, single-blind period precedes the 8-week randomized treatment period and an optional 18-week, double-blind extension period follows the randomized treatment period. A Safety Follow up Visit is scheduled 1 week after the acute and extension period, or early termination. Escitalopram, a selective serotonin reuptake inhibitor (SSRI), an approved treatment for MDD, is chosen as a positive control agent in this study. The dose of 10 mg is within the approved dose range with no need for dose adjustment in elderly patients. This trial is designed to formally compare the efficacy, safety, and tolerability of SR58611A to placebo. Escitalopram is used as a positive control.

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria:

* 1. Out-patients, 18 year and older.
* 2. Major Depressive Disorder (MDD) with a recurrentMajor Depressive Episode (MDE) according to DSMIV-TR criteria
* 3. Duration of current episode is at least of 6 weeksunless severity of symptoms justifies shorter duration.
* 4. Patients have been treated or hospitalized for aprevious episode, or a previous episode requiredantidepressant treatment(s) at the recommended doselevel for a continuous total duration of at least 2months.

Exclusion Criteria:

Main exclusion criteria:

* 1. Patients at immediate risk for suicidal behavior
* 2. Patients with a MDE with psychotic features, catatonic features, seasonal pattern or postpartum onset
* 3. The duration of the current depressive episode is greater than 2 years
* 4. Patients whose current depressive episode is secondary to a general medical condition
* 5. Patients with a lifetime history of (1) bipolar disorder, (2) psychotic disorder, (3) antisocial personality disorder
* 6. Patients who have received non-pharmacologic, somatic treatments for psychiatric disease
* 7. Patients who have initiated, stopped, or changed the frequency or nature of psychotherapy within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Depression Rating Scale (HAM-D) total score

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impression (CGI) and MADRS Severity of Illness score
Safety assessments

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Laval, Canada

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com